CLINICAL TRIAL: NCT05231135
Title: Characteristics, Treatment and Outcomes of HIV-infected Patients With Malignant Lymphoma: A Registry Study of the European Hematology Association (EHA) Lymphoma Group
Brief Title: A Registry Study on HIV-related Lymphoma
Status: Recruiting | Type: Observational
Sponsor: Rotkreuzklinikum München gGmbH (Other)
Responsible Party: Principal Investigator, Prof. Marcus Hentrich, Head of the Department of Hematology and Oncology, Rotkreuzklinikum München gGmbH
Other Study IDs: IN03/0121
Record Dates: First submitted 2022-01-05; First posted 2022-02-09 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: AIDS Related Lymphoma; HIV Related Lymphoma
Keywords: Malignant lymphoma; HIV-related lymphoma; HIV-associated Hodgkin lymphoma
MeSH Terms: conditions — Lymphoma, AIDS-Related; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective und prospective registry on HIV-associated lymphoma. Data on characteristics, type and toxicity of treatment and outcome of patients with HIV-lymphoma will be collected.

DETAILED DESCRIPTION:
To study characteristics, treatment approaches and outcome of HIV-infected patients with malignant lymphoma in the combination antiretroviral therapy (cART) era. HIV-infected persons diagnosed with non-Hodgkin lymphoma or Hodgkin lymphoma will be included. The choice of treatment is not specified by the registry study. However, the type of antineoplastic treatment should follow national or international recommendations and guidelines. Data will be pseudonymized by the data manager of the treating institution. Central data management is located at Red Cross Hospital Munich, Germany.

ELIGIBILITY:
Inclusion Criteria:

* Histology or cytology proven non-Hodgkin lymphoma or Hodgkin lymphoma
* HIV-infection at time of lymphoma diagnosis
* Lymphoma diagnosis since 01.01.2010
* Adult patients ≥ 18 years
* Written informed consent

Exclusion Criteria:

* HIV-diagnosis > 3 months after the diagnosis of malignant lymphoma
* Non-Compliance or lack of opportunity for follow-up (for the prospective part of the study)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unselected cohort of adults with HIV-lymphoma
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
2-year overall survival (OS) | 2 years
  OS measured from the date of diagnosis to last follow-up or to death from any cause.
2-year progression-free survival (PFS) | 2 years
  PFS calculated from the date of diagnosis to the time of progression, relapse, or death.

SECONDARY OUTCOMES:
Incidence of relapse (IR) | 5 years
  Based on establised response criteria, e.g. Chesson et al. JCO 2014
Non-relapse mortality (NRM) | 5 years
  Deaths unrelated to lymphoma
5-year overall survival (OS) | 5 years
  OS measured from the date of diagnosis to last follow-up or to death from any cause.
5-year progression-free survival (PFS) | 5 years
  PFS calculated from the date of diagnosis to the time of progression, relapse, or death.

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Hentrich, MD, Study Chair — Rotkreuzklinikum München
Locations (6):
- Germany (2):
  - Red Cross Hospital Munich, Munich, Select One Option
  - University Hospital Cologne, Cologne
- Amsterdam University Medical Centers, Amsterdam, Netherlands
- Spain (2):
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
- University Hospital of Wales, Cardiff, United Kingdom